CLINICAL TRIAL: NCT05392439
Title: The Efficacy and Mechanisms of Transcutaneous Auricular Vagus Nerve Stimulation on Abdominal Pain and Other Symptoms in Patients With Constipation-predominant Irritable Bowel Syndrome
Brief Title: Effect of taVNS on Abdominal Pain and Other Symptoms in Constipation-predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji University (Other)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Shi, Junior Physician, Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-006
Record Dates: First submitted 2022-05-21; First posted 2022-05-26 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome; Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS treatment (Experimental): The taVNS treatment is performed at auricular cymba concha. The stimulation parameters are set as follows: train on-time of 2 seconds and off-time of a 3-second pulse width of 0.5 ms, pulse frequency of 25 Hz, and amplitude of 0-2 milliamp (at the maximum level tolerated by the subject).
  Interventions: Device: taVNS
- sham-taVNS treatment (Sham Comparator): Sham-taVNS is performed with the same parameters as taVNS except that electrical stimulation is applied at the elbow area.
  Interventions: Device: sham-taVNS

INTERVENTIONS:
Device: taVNS — transcutaneous auricular vagal nerve stimulation
  Arms: taVNS treatment
Device: sham-taVNS — transcutaneous stimulation at the elbow area
  Arms: sham-taVNS treatment

SUMMARY:
This study aims to investigate the effects and possible mechanisms of transcutaneous auricular vagal nerve stimulation (taVNS) on abdominal pain and other symptoms in patients with IBS-C.

DETAILED DESCRIPTION:
This study is designed as an early-feasibility, single-center, single-blinded, randomized controlled trial (RCT), in which subjects are consented, undergo a baseline assessment, and receive taVNS or sham-taVNS treatment twice a day (8 a.m. and 8 p.m.) for 30 minutes each time for a period of 4 weeks. The taVNS and sham-taVNS treatment was applied using the commercially-available Transcutaneous Electrical Applicator device (Model SNM-FDC01, Ningbo MedKinetic Medical Device Co., Ltd.) with the skin electrodes placed bilaterally on auricular concha. The patients are requested to score the abdominal pain (using VAS) and complete BSFS, IBS-SSS, IBS-QOL, SAS, and SDS forms every week and fill out the bowel diary during taVNS or sham-taVNS. Emergency medications (Macrogol 4000 and pinaverium) are permitted for use when the patient cannot tolerate symptoms of constipation and abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

1. willing to sign a written informed consent form
2. met the Rome IV diagnostic criteria for IBS-C

Exclusion Criteria:

1. history of previous abdominal surgery (other than appendectomy)
2. presence of carcinoma
3. any organic diseases causing constipation or neurologic diseases such as multiple sclerosis, rachischisis, Parkinson's disease, or spinal cord injury
4. taking antidepressant agents including tricyclic antidepressants and selective serotonin reuptake inhibitors
5. serious concomitant disease of the heart, liver, kidney, or diabetes
6. pregnancy or lactation
7. participating in another trial or enrolled in a trial during the past month
8. allergic reaction to surface electrodes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Change in аbdominal pain between sham and active taVNS | 4 weeks
  Weekly average of daily patient-assessed abdominal pain using the visual analog scale (VAS). VAS ranges from 0 to 10, with 0 indicating no abdominal pain and 10 indicating the maximal pain. Efficacy is evaluated as an improvement of ≥ 30%.

SECONDARY OUTCOMES:
Change in IBS symptom severity scale (IBS-SSS) between sham and active taVNS | 4 weeks
  Questionnaire consists of 5 questions (abdominal pain intensity, abdominal pain frequency, abdominal distension degree, defecation satisfaction, and interference with quality of life), with a total score of 500 points and a higher score indicating a worse condition. Scores < 175 represent mild IBS symptoms, scores 175-300 represent moderate severity, and scores > 300 represent severe IBS.
Change in IBS quality of life (IBS-QOL) between sham and active taVNS | 4 weeks
  Questionnaire is composed of 8 dimensions (dysphoria, interference with activity, body image, health concerns, food avoidance, social reaction, sex, and relationships), with 34 items assessing the degree to which IBS interferes with the patient's quality of life. Each item is evaluated on a 5-point Likert scale. The total score ranges from 34 to 170 and higher scores indicate better quality of life.
Change in Bristol stool form scale (BSFS) between sham and active taVNS | 4 weeks
  The scale has 7 points according to stool type, from the hardest (1) to the softest (7). The lower the score, the more severe is constipation.
Change in Self-Rating Anxiety Scale (SAS) score between sham and active taVNS | 4 weeks
  SAS questionnaire has 20 items to assess physical and psychological symptoms, using a 4-point Likert scale ranging from 1 (none, or a little of the time) to 4 (most, or all of the time), with a total score ranging from 20 to 80. SAS scores below 50 indicate no anxiety, from 50 to 59 - mild anxiety, from 60 to 69 - moderate anxiety, 70 and above - severe anxiety.
Change in Self-Rating Depression Scale (SDS) score between sham and active taVNS | 4 weeks
  SDS questionnaire has 20 items to assess physical and psychological symptoms, using a 4-point Likert scale ranging from 1 (none, or a little of the time) to 4 (most, or all of the time), with a total score ranging from 20 to 80. SDS scores below 50 indicate no depression, from 50 to 59 - mild depression, from 60 to 69 - moderate depression, 70 and above - severe depression.
Change in complete spontaneous bowel movements per week between sham and active taVNS | 4 weeks
  Number of bowel movements that occur without use of any medication or other methods to assist defecation and with a feeling of complete evacuation

OTHER OUTCOMES:
Change in autonomic function assessed by the spectral parameters of heart rate variability between sham and active stimulation | 4 weeks
  Heart rate variability parameters are calculated using spectral analysis of R-R intervals in electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, China

REFERENCES:
- [Result] Shi X, Hu Y, Zhang B, Li W, Chen JD, Liu F. Ameliorating effects and mechanisms of transcutaneous auricular vagal nerve stimulation on abdominal pain and constipation. JCI Insight. 2021 Jul 22;6(14):e150052. doi: 10.1172/jci.insight.150052. PMID 34138761

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/39/NCT05392439/Prot_SAP_000.pdf